CLINICAL TRIAL: NCT02155647
Title: A Phase II, Open-Label, Multicenter Trial to Investigate the Clinical Activity and Safety of Avelumab (MSB0010718C) in Subjects With Merkel Cell Carcinoma
Brief Title: Avelumab in Participants With Merkel Cell Carcinoma (JAVELIN Merkel 200)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100070-003; 2014-000445-79 (EudraCT Number)
Record Dates: First submitted 2014-06-02; First posted 2014-06-04 (Estimated); Results first posted 2020-07-22 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Merkel Cell
Keywords: Carcinoma, Merkel Cell; MSB0010718C; avelumab; Bavencio; anti PD-L1; JAVELIN Merkel 200
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Part A: Avelumab (Experimental): Participants with metastatic Merkel cell carcinoma (MCC) after failing first-line chemotherapy received Avelumab at a dose of 10 milligram per kilogram (mg/kg) as 1-hour intravenous infusion once every 2 weeks until therapeutic failure, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the trial or investigational medicinal product occurs.
  Interventions: Drug: Avelumab
- Part B: Avelumab (Experimental): Participants received Avelumab as first-line treatment for metastatic or distally recurrent MCC at a dose of 10 mg/kg as 1-hour intravenous infusion once every 2 weeks until therapeutic failure, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the trial or investigational medicinal product occurs.
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Avelumab was administered at a dose of 10 milligram per kilogram (mg/kg) as 1-hour intravenous infusion once every 2 weeks until therapeutic failure, significant clinical deterioration, unacceptable toxicity, or any criterion for withdrawal from the trial or investigational medicinal product occurs.
  Other Names: anti-PD-L1; MSB0010718C

SUMMARY:
This is a multicenter, international, single-arm, open-label, Phase 2 trial to evaluate the efficacy and safety of avelumab in participants with metastatic Merkel cell carcinoma (MCC).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Age 18 years and above
* Histologically proven MCC
* Participants must have received at least 1 line of chemotherapy for metastatic MCC and must have progressed after the most recent line of chemotherapy
* For Part B - Participants must not have received any prior systemic treatment for metastatic MCC. Prior chemotherapy treatment in the adjuvant setting (no clinically detectable disease; no metastatic disease) is allowable if the end of treatment occurred at least 6 months prior to study start)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Disease must be measurable with at least 1 uni-dimensional measurable lesion by RECIST Version 1.1 (including skin lesions)
* Adequate hematological, hepatic and renal function (renal function considered adequate as per protocol definition)
* Highly effective contraception for both male and female participants, if the risk of conception exists
* Fresh Biopsy or Archival Tumor Tissue
* Estimated life expectancy of more than 12 weeks

Exclusion Criteria:

* Participation in another interventional clinical trial within the past 30 days (participation in observational studies is permitted)
* Concurrent treatment with a non permitted drug
* Prior therapy with any antibody/drug targeting T-cell coregulatory proteins (immune checkpoints) such as antiprogrammed death 1 (PD-1), anti-PD-L1, or anticytotoxic T-lymphocyte antigen-4 (CTLA-4) antibody; for Part B, the Investigator must consult with the Medical Monitor and consider other co-regulatory targets such as 4-1BB
* Concurrent anticancer treatment (for example, cytoreductive therapy, radiotherapy [with the exception of palliative bone-directed radiotherapy, or radiotherapy administered on non-target superficial lesions], immune therapy, or cytokine therapy except for erythropoietin). Radiotherapy administered to superficial lesions is not allowed if such lesions are considered target lesions in the efficacy evaluation or may influence the efficacy evaluation of the investigational agent
* Major surgery for any reason, except diagnostic biopsy, within 4 weeks and/or if the participant has not fully recovered from the surgery within 4 weeks
* Concurrent systemic therapy with steroids or other immunosuppressive agents, or use of any investigational drug within 28 days before the start of trial treatment. Short-term administration of systemic steroids (that is, for allergic reactions or the management of immune-related adverse events [irAE]) while on study is allowed. Also, participants requiring hormone replacement with corticosteroids for adrenal insufficiency are eligible if the steroids are administered only for the purpose of hormonal replacement and at doses <= 10 mg or equivalent prednisone per day. Note: Participants receiving bisphosphonate or denosumab are eligible.
* Participants with active central nervous system (CNS) metastases are excluded. Participants with a history of treated CNS metastases (by surgery or radiation therapy) are not eligible unless they have fully recovered from treatment, demonstrated no progression for at least 2 months, and do not require continued steroid therapy
* Previous malignant disease (other than MCC) within the last 5 years with the exception of basal or squamous cell carcinoma of the skin and for Part A cervical carcinoma in situ or for Part B carcinoma in situ (skin, bladder, cervical, colorectal, breast or low grade prostatic intraepithelial neoplasia or Grade 1 prostate cancer)
* Prior organ transplantation, including allogeneic stem-cell transplantation
* Part A: Known history of testing positive for HIV or known acquired immunodeficiency syndrome (AIDS) or any positive test for hepatitis B virus or hepatitis C virus indicating acute or chronic infection. For Part B, known history of testing positive for HIV or known AIDS in consultation with the Medical Monitor or HBV or HCV infection at screening (positive HBV surface antigen or HCV RNA if anti- HCV antibody screening test positive).
* Active or history of any autoimmune disease (except for participants with vitiligo) or immunodeficiencies that required treatment with systemic immunosuppressive drugs
* Known severe hypersensitivity reactions to monoclonal antibodies (Grade greater than or equal to (>=) 3 NCI CTCAE v 4.0), any history of anaphylaxis, or uncontrolled asthma (that is, 3 or more features of partially controlled asthma)
* Persisting toxicity related to prior therapy Grade > 1 NCI-CTCAE v 4.0; however, sensory neuropathy Grade <= 2 is acceptable 14. Pregnancy or lactation
* Known alcohol or drug abuse
* Clinically significant (that is, active) cardiovascular disease: cerebral vascular accident / stroke (< 6 months prior to enrollment), myocardial infarction (< 6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class >= II), or serious cardiac arrhythmia requiring medication
* All other significant diseases (for example, inflammatory bowel disease), which, in the opinion of the Investigator, might impair the participant's tolerance of trial treatment
* Any psychiatric condition that would prohibit the understanding or rendering of informed consent
* Legal incapacity or limited legal capacity
* Non oncology vaccine therapies for prevention of infectious disease (for example, seasonal flu vaccine, human papilloma virus vaccine) within 4 weeks of trial drug administration. Vaccination while on trial is also prohibited except for administration of inactivated vaccines (for example, inactivated seasonal influenza vaccine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Actual)
Dates: Start 2014-07-03 (Actual); Primary Completion 2019-05-02 (Actual); Study Completion 2023-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (61):
- United States (14):
  - UCLA Medical Center, Los Angeles, California
  - The Angeles Clinic and Research Institute - West LA, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - H. Lee Moffitt Cancer Center and Research Institute, Inc, Tampa, Florida
  - National Cancer Institute, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Mount Sinai, New York, New York
  - Peggy & Charles Stephenson Oklahoma Cancer Center, Oklahoma City, Oklahoma
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Washington - Seattle Cancer Care Alliance, Seattle, Washington
- Australia (6):
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Tasman Oncology Research Ltd, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - St John of God Subiaco Hospital, Perth, Western Australia
- France (14):
  - CHU Nice - Hopital de l Archet 2, Nice, Alpes Maritimes
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - CHU Nantes - Hôtel Dieu, Nantes, Loire Atlantique
  - Hopital Claude Huriez - CHU Lille, Lille, Nord
  - Hôpital Saint-Louis, Paris, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhone
  - Institut Gustave Roussy, Villejuif, Val De Marne
  - Groupe Hospitalier Saint André - Hôpital Saint André, Bordeaux
  - Hôpital Ambroise Paré - Boulogne-Billancourt, Boulogne-Billancourt
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours
  - CHU de Dijon - Hopital du Bocage, Dijon
  - CHU de Grenoble - Hôpital A Michallon, Grenoble
  - CHU de Limoges - Hôpital Dupuytren, Limoges
- Germany (11):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Klinikum der Johann Wolfgang Goethe-Universitaet, Frankfurt am Main, Hesse
  - St. Josef-Hospital Universitaetsklinikum, Bochum, North Rhine-Westphalia
  - Universitaetsklinikum Koeln, Cologne, North Rhine-Westphalia
  - Universitaetsklinikum Essen, Essen, North Rhine-Westphalia
  - Fachklinik Hornheide, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitaetsklinikum Schleswig-Holstein - Klinik fuer Allgemeine Innere Medizin, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Schleswig Holstein - Campus Luebeck, Lübeck, Schleswig-Holstein
  - Helios Klinikum Erfurt, Erfurt, Thuringia
  - Charite Universitaetsmedizin Berlin - Campus Charite Mitte, Berlin
- Italy (9):
  - Fondazione del Piemonte per l'Oncologia IRCC Candiolo, Candiolo, Torino
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - IEO Istituto Europeo di Oncologia, Milan
  - Istituto Nazionale Tumori Fondazione G.Pascale, Napoli
  - IOV - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliera di Perugia Ospedale S. Maria della Misericordia, Perugia
  - Arcispedale S. Maria Nuova Azienda Ospedaliera di Reggio Emilia, Reggio Emilia
  - Istituto Nazionale Tumori Regina Elena IRCCS, Roma
  - A.O.U. Senese Policlinico Santa Maria alle Scotte, Siena
- Japan (2):
  - Shizuoka Cancer Center, Shizuoka, Shizuoka
  - National Cancer Center Hospital, Chūōku
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital General Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Per company policy, following approval of a new product or a new indication for an approved product in both the EU and the US, EMD Serono will share study protocols, anonymized patient level and study level data and redacted clinical study reports from clinical trials in patients with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website https://www.emdgroup.com/en/research/our-approach-to-research-and-development/healthcare/clinical-trials/commitment-responsible-data-sharing.html
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Within six months after the approval of a new product or a new indication for an approved product in both the United States and the European Union
Access Criteria: Qualified scientific and medical researchers can request the data. Such requests must be submitted in writing to the company's portal and will be internally reviewed regarding criteria for researchers' qualification and legitimacy of the research proposal.
URL: http://bit.ly/IPD21

REFERENCES:
- [Result] Kaufman HL, Russell J, Hamid O, Bhatia S, Terheyden P, D'Angelo SP, Shih KC, Lebbe C, Linette GP, Milella M, Brownell I, Lewis KD, Lorch JH, Chin K, Mahnke L, von Heydebreck A, Cuillerot JM, Nghiem P. Avelumab in patients with chemotherapy-refractory metastatic Merkel cell carcinoma: a multicentre, single-group, open-label, phase 2 trial. Lancet Oncol. 2016 Oct;17(10):1374-1385. doi: 10.1016/S1470-2045(16)30364-3. Epub 2016 Sep 1. PMID 27592805
- [Result] Kaufman HL, Russell JS, Hamid O, Bhatia S, Terheyden P, D'Angelo SP, Shih KC, Lebbe C, Milella M, Brownell I, Lewis KD, Lorch JH, von Heydebreck A, Hennessy M, Nghiem P. Updated efficacy of avelumab in patients with previously treated metastatic Merkel cell carcinoma after >/=1 year of follow-up: JAVELIN Merkel 200, a phase 2 clinical trial. J Immunother Cancer. 2018 Jan 19;6(1):7. doi: 10.1186/s40425-017-0310-x. PMID 29347993
- [Result] D'Angelo SP, Russell J, Lebbe C, Chmielowski B, Gambichler T, Grob JJ, Kiecker F, Rabinowits G, Terheyden P, Zwiener I, Bajars M, Hennessy M, Kaufman HL. Efficacy and Safety of First-line Avelumab Treatment in Patients With Stage IV Metastatic Merkel Cell Carcinoma: A Preplanned Interim Analysis of a Clinical Trial. JAMA Oncol. 2018 Sep 1;4(9):e180077. doi: 10.1001/jamaoncol.2018.0077. Epub 2018 Sep 13. PMID 29566106
- [Result] D'Angelo SP, Bhatia S, Brohl AS, Hamid O, Mehnert JM, Terheyden P, Shih KC, Brownell I, Lebbe C, Lewis KD, Linette GP, Milella M, Georges S, Shah P, Ellers-Lenz B, Bajars M, Guzel G, Nghiem PT. Avelumab in patients with previously treated metastatic Merkel cell carcinoma: long-term data and biomarker analyses from the single-arm phase 2 JAVELIN Merkel 200 trial. J Immunother Cancer. 2020 May;8(1):e000674. doi: 10.1136/jitc-2020-000674. PMID 32414862
- [Result] Lambert J, Marrel A, D'Angelo SP, Burgess MA, Chmielowski B, Fazio N, Gambichler T, Grob JJ, Lebbe C, Robert C, Russell J, Guzel G, Bharmal M. Patient Experiences with Avelumab in Treatment-Naive Metastatic Merkel Cell Carcinoma: Longitudinal Qualitative Interview Findings from JAVELIN Merkel 200, a Registrational Clinical Trial. Patient. 2020 Aug;13(4):457-467. doi: 10.1007/s40271-020-00428-5. PMID 32472503
- [Result] Kaufman HL, Dias Barbosa C, Guillemin I, Lambert J, Mahnke L, Bharmal M. Living with Merkel Cell Carcinoma (MCC): Development of a Conceptual Model of MCC Based on Patient Experiences. Patient. 2018 Aug;11(4):439-449. doi: 10.1007/s40271-018-0301-0. PMID 29512061
- [Result] Bharmal M, Fofana F, Barbosa CD, Williams P, Mahnke L, Marrel A, Schlichting M. Psychometric properties of the FACT-M questionnaire in patients with Merkel cell carcinoma. Health Qual Life Outcomes. 2017 Dec 22;15(1):247. doi: 10.1186/s12955-017-0815-5. PMID 29273043
- [Result] Kelly K, Manitz J, Patel MR, D'Angelo SP, Apolo AB, Rajan A, Kasturi V, Speit I, Bajars M, Warth J, Gulley JL. Efficacy and immune-related adverse event associations in avelumab-treated patients. J Immunother Cancer. 2020 Nov;8(2):e001427. doi: 10.1136/jitc-2020-001427. PMID 33219092
- [Result] Bharmal M, Nolte S, Lebbe C, Mortier L, Brohl AS, Fazio N, Grob JJ, Pusceddu S, Hanna GJ, Hassel JC, Kiecker F, Ellers-Lenz B, Bajars M, Guzel G, Nghiem P, Hunger M, Schlichting M, Henry-Szatkowski M, D'Angelo SP. Health-related quality of life trajectory of treatment-naive patients with Merkel cell carcinoma receiving avelumab. Future Oncol. 2020 Sep;16(27):2089-2099. doi: 10.2217/fon-2020-0426. Epub 2020 Sep 17. PMID 32938212
- [Derived] Grisic AM, Xiong W, Tanneau L, Jonsson S, Friberg LE, Karlsson MO, Dai H, Zheng J, Girard P, Khandelwal A. Model-Based Characterization of the Bidirectional Interaction Between Pharmacokinetics and Tumor Growth Dynamics in Patients with Metastatic Merkel Cell Carcinoma Treated with Avelumab. Clin Cancer Res. 2022 Apr 1;28(7):1363-1371. doi: 10.1158/1078-0432.CCR-21-2662. PMID 34921021
- [Derived] D'Angelo SP, Lebbe C, Mortier L, Brohl AS, Fazio N, Grob JJ, Prinzi N, Hanna GJ, Hassel JC, Kiecker F, Georges S, Ellers-Lenz B, Shah P, Guzel G, Nghiem P. First-line avelumab in a cohort of 116 patients with metastatic Merkel cell carcinoma (JAVELIN Merkel 200): primary and biomarker analyses of a phase II study. J Immunother Cancer. 2021 Jul;9(7):e002646. doi: 10.1136/jitc-2021-002646. PMID 34301810
- [Derived] Bharmal M, Nolte S, Henry-Szatkowski M, Hennessy M, Schlichting M. Update on the psychometric properties and minimal important difference (MID) thresholds of the FACT-M questionnaire for use in treatment-naive and previously treated patients with metastatic Merkel cell carcinoma. Health Qual Life Outcomes. 2020 May 19;18(1):145. doi: 10.1186/s12955-020-01402-3. PMID 32430019
- [Derived] Bullement A, Willis A, Amin A, Schlichting M, Hatswell AJ, Bharmal M. Evaluation of survival extrapolation in immuno-oncology using multiple pre-planned data cuts: learnings to aid in model selection. BMC Med Res Methodol. 2020 May 6;20(1):103. doi: 10.1186/s12874-020-00997-x. PMID 32375680
- [Derived] Novakovic AM, Wilkins JJ, Dai H, Wade JR, Neuteboom B, Brar S, Bello CL, Girard P, Khandelwal A. Changing Body Weight-Based Dosing to a Flat Dose for Avelumab in Metastatic Merkel Cell and Advanced Urothelial Carcinoma. Clin Pharmacol Ther. 2020 Mar;107(3):588-596. doi: 10.1002/cpt.1645. Epub 2019 Nov 18. PMID 31553054
- [Derived] Bharmal M, Guillemin I, Marrel A, Arnould B, Lambert J, Hennessy M, Fofana F. How to address the challenges of evaluating treatment benefits-risks in rare diseases? A convergent mixed methods approach applied within a Merkel cell carcinoma phase 2 clinical trial. Orphanet J Rare Dis. 2018 Jun 18;13(1):95. doi: 10.1186/s13023-018-0835-1. PMID 29914528
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=100070-003
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 88 participants were enrolled in Part A of the study and a total of 116 participants were enrolled in Part B of the study. Participants enrolled in Part A were not eligible for enrollment in Part B.
Period: Overall Study
Arm/Group | Part A: Avelumab | Part B: Avelumab
Started | 88 | 116
Completed | 88 | 116
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part A: Avelumab | Part B: Avelumab | Total
Number analyzed (Participants) | 88 | 116 | 204
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 66 | 94 | 160
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 35 | 58
  Male | 65 | 81 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 29 | 33
  Not Hispanic or Latino | 58 | 75 | 133
  Unknown or Not Reported | 26 | 12 | 38
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 81 | 75 | 156
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 36 | 40

OUTCOME MEASURES:

1. Primary Outcome: Part A: Number of Participants With Confirmed Best Overall Response (BOR) as Per Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
Description: Confirmed BOR was determined according to RECIST 1.1and as adjudicated by an Independent Endpoint Review Committee(IERC) and defined as best response of any of complete response (CR), partial response(PR), stable disease(SD) and progressive disease(PD) recorded from date of randomization until disease progression/recurrence(taking smallest measurement recorded since start of treatment as reference). CR:Disappearance of all evidence of target/non-target lesions. PR:At least 30%reduction from baseline in sum of longest diameter(SLD) of all lesions. SD:Neither sufficient increase to qualify for PD nor sufficient shrinkage to qualify for PR. PD:at least a20% increase in SLD, taking as reference smallest SLD recorded from baseline/appearance of 1or more new lesions and unequivocal progression of non-target lesions. CR or PR must be confirmed by a subsequent tumor assessment preferably at next scheduled 6-weekly assessment, but no sooner than 5 weeks after initial documentation of CR or PR.
Time Frame: Up to 113 weeks
Population: Intent-to-Treat analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Participants
  Complete Response | 10
  Partial Response | 19
  Stable Disease | 9
  Non-complete Response/ Non-progressive Disease | 0
  Progressive Disease | 32
  Not evaluable | 18

2. Primary Outcome: Part B: Durable Response Rate (DRR)
Description: Durable response is defined as an objective response (confirmed complete response [CR] or confirmed Partial response [PR]) according to Response Evaluation Criteria in Solid Tumors version (RECIST) 1.1, determined by the Independent Endpoint Review Committee (IERC), with a duration of at least 6 months. The DRR was determined as the percentage of participants with an objective response in terms of CR or PR according to RECIST 1.1, as determined by the IERC, with a duration of at least 6 months. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions.
Time Frame: Up to 161 weeks
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
Percentage of participants | 30.2 [22.0 to 39.4]

3. Secondary Outcome: Part A: Duration of Response According to Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
Description: The duration of response as determined from IERC tumor assessment was calculated for each participant with a confirmed response (CR or PR) as the time from first observation of response until first observation of documented disease progression or death when death occurs within 12 weeks of the last tumor assessment, whichever occurs first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Results were calculated based on Kaplan-Meier estimates.
Time Frame: Up to 325 weeks
Population: Intent-to-Treat analysis set included all participants who received at least 1 dose of study treatment. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 29
Months | 40.5 [2.8 to 41.5]

4. Secondary Outcome: Part A: Progression-Free Survival (PFS) Time According to Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
Description: The PFS time (based on IERC tumor assessments), according to the RECIST 1.1, was defined as the time from first administration of study treatment until first observation of PD or death when death occurred within 12 weeks of the last tumor assessment or first administration of study treatment (whichever was later). PFS time (in months) was defined as: (date of PD or death - date of the first dose of study treatment + 1)/30.4375 (months). PD was defined as at least a 20% increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions and unequivocal progression of non-target lesions.
Time Frame: Up to 325 weeks
Population: Intent-to-Treat analysis set included all participants who received at least 1 dose of study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Months | 2.7 [0.03 to 45.6]

5. Secondary Outcome: Part A: Number of Participants With Treatment-Related (TR) Treatment-Emergent Adverse Events (TEAEs), Treatment-Related Serious TEAEs and Treatment-Related TEAEs Leading to Death
Description: Related Adverse events (AE) were defined according to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI-CTCAE) as adverse events with relationship to study treatment reported by the investigator. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Treatment-emergent are events between first dose of study drug that were absent before treatment or that worsened relative to pre-treatment state up to 30 days after last administration. TEAEs included both Serious TEAEs and non-serious TEAEs. Related TEAEs are defined as events with a relationship of missing, unknown, or yes.
Time Frame: Up to 325 weeks
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Participants
  Participants with TR-TEAEs | 68
  Participants with TR-Serious-TEAEs | 9
  Participants with TR-TEAEs leading to Death | 0

6. Secondary Outcome: Part A: Number of Participants With Clinically Significant Abnormalities in Laboratory Values Reported as Treatment Emergent Adverse Events (TEAEs)
Description: The laboratory measurements included hematology, liver function and blood chemistry. Number of participants with clinically significant abnormalities with Grade greater than or equals to (>=) 3 in laboratory values reported as TEAEs were reported. Clinically Significance was decided by investigator.
Time Frame: Up to 325 weeks
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Participants
  Anemia | 9
  Lymphocyte count decreased | 18
  Neutrophil count decreased | 1
  Platelet count decreased | 1
  White blood cell count decreased | 1
  Hypoalbuminemia | 2
  Alkaline phosphatase increased | 1
  Alanine aminotransferase increased | 3
  Serum amylase increased | 1
  Aspartate aminotransferase increased | 1
  Blood bilirubin increased | 1
  Cholesterol high | 1
  Creatine phosphokinase increased | 1
  Creatinine increased | 2
  Chronic kidney disease | 3
  Gamma-glutamyltransferase increased | 6
  Hyperglycemia | 7
  Hypoglycemia | 1
  Hyperkalemia | 1
  Hypokalemia | 2
  Lipase increased | 4
  Hypermagnesemia | 1
  Hypophosphatemia | 3
  Hyponatremia | 11
  Hypertriglyceridemia | 1

7. Secondary Outcome: Part A: Number of Participants With Clinically Significant Abnormalities in Vital Signs Reported as Treatment Emergent Adverse Events (TEAEs)
Description: Vital signs including body temperature, body weight, respiratory rate, heart rate (after 5-minute rest), and arterial blood pressure (after 5-minute rest) were evaluated. Number of participants with clinically significant abnormalities in Vital Signs reported as TEAEs. Clinically Significance was decided by investigator.
Time Frame: Up to 325 weeks
Population: Safety analysis set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Participants
  Body temperature Increased | 0
  Weight Increased | 57
  Weight Decreased | 54
  Increased Heart Rate | 83
  Decreased Heart Rate | 84
  Increased Systolic Blood Pressure | 84
  Decreased Systolic Blood Pressure | 84
  Increased Diastolic Blood Pressure | 84
  Decreased Diastolic Blood Pressure | 84
  Increased Respiratory Rate | 81
  Decreased Respiratory Rate | 81

8. Secondary Outcome: Part A: Number of Participants With Clinically Significant Abnormalities in Electrocardiogram (ECG)
Description: A 12-lead ECG was recorded after the participant has been in a supine position breathing quietly for 5 minutes. The ECG results was used to evaluate the heart rate, atrial ventricular conduction, PR interval, QRS, QTcF and QTcB. Number of participants with clinical significant abnormalities in ECG parameter reported here. Clinically Significance was decided by investigator.
Time Frame: Up to 325 weeks
Population: Safety analysis set included all participants who received at least 1 dose of study treatment. Here "Number of participants analyzed" signifies those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 81
Participants
  PR interval >= 220 ms | 16
  QRS >= 120 ms | 12
  QTcF > 30 ms and <= 60 ms | 20
  QTcF > 60 ms | 1
  QTcB > 30 ms and <= 60 ms | 25
  QTcB > 60 ms | 2
  Heart rate <= 50 bpm | 3
  Heart rate >= 120 bpm | 2

9. Secondary Outcome: Part A: Interim Analysis: Overall Survival (OS) Time
Description: The OS time was defined as the time from first administration of trial treatment until death. The OS time was analyzed using the Kaplan-Meier method.
Time Frame: Up to 87 weeks (Data reported are per pre-specified interim analysis with a data cut-off date of 3 Mar 2016)
Population: Intent-to-Treat analysis set included all participants who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Months | 11.3 [7.5 to 14.0]

10. Secondary Outcome: Part A: Final Analysis: Overall Survival (OS) Time
Description: as for outcome 9
Time Frame: Time from first administration of trial treatment until death (Up to 325 weeks)
Population: Intent-to-Treat analysis set included all participants who received at least 1 dose of study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
months | 12.6 [0.4 to 71.9]

11. Secondary Outcome: Part A: Participant's Response Status According to Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1 at 6 and 12 Months
Description: The response status at 6 and 12 months after start of trial treatment according to RECIST 1.1 (as determined by the IERC) was determined. A participant was considered to be in response at the given timepoint (6 or 12 months after the start of the participant's treatment) if the participant had a documented response (PR or CR) prior to that timepoint, and neither died nor experienced disease progression according to the RECIST 1.1 nor was lost to follow-up up to the given timepoint. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Percentage of participants in response and not in response according to RECIST1.1 at 6 and 12 months were reported.
Time Frame: At Month 6 and 12
Population: Intent-to-Treat analysis set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Percentage of participants
  In-response at Month 6 | 30.7
  In-response at Month 12 | 20.7
  Not in-response at Month 6 | 69.3
  Not In-response at Month 12 | 79.3

12. Secondary Outcome: Part A: Number of Participants With Positive Treatment Emergent Anti-Avelumab Antibodies
Description: Serum samples were analyzed by a validated electrochemiluminesce immunoassay to detect the presence of anti-avelumab antibodies. Samples that screened positive were subsequently tested in a confirmatory assay. Those confirmed positive were titered for a quasi-quantitative result. Number of participants with positive treatment emergent anti-Avelumab antibodies were reported. Participants not positive prior to treatment with avelumab and with at least one positive result in the human-Antihuman Antibodies assay were characterized as treatment-emergent.
Time Frame: Up to 80 weeks
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 82
Participants | 3

13. Secondary Outcome: Part A: Serum Concentration at End of Infusion (CEOI) of Avelumab
Description: Serum concentration at end of infusion (CEOI) of Avelumab is reported.
Time Frame: Day 1, 43, 85, 169, 253, 337 and 421
Population: Pharmacokinetic analysis set consists of all participants who received at least 1 dose of avelumab, and provide at least 1 measurable post-dose concentration. Here "Number analyzed" signifies those participants who were evaluable at specified timepoints
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Micrograms per milliliter
  Day 1: number analyzed (Participants) | 59
  Day 1 | 252 (129)
  Day 43: number analyzed (Participants) | 48
  Day 43 | 266 (74.2)
  Day 85: number analyzed (Participants) | 30
  Day 85 | 274 (57.7)
  Day 169: number analyzed (Participants) | 23
  Day 169 | 315 (65.0)
  Day 253: number analyzed (Participants) | 15
  Day 253 | 318 (70.1)
  Day 337: number analyzed (Participants) | 6
  Day 337 | 373 (48.3)
  Day 421: number analyzed (Participants) | 4
  Day 421 | 453 (71.5)

14. Secondary Outcome: Part A: Minimum Serum Post-dose (Ctrough) Concentration of Aveluamb
Description: Minimum serum post-dose (Ctrough) concentration of avelumab was reported.
Time Frame: Day 15, 29, 43, 57, 71, 85, 99, 169, 211, 253, 337 and 421
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Micrograms per milliliter
Arm/Group | Part A: Avelumab
Number analyzed (Participants) | 88
Micrograms per milliliter
  Day 15: number analyzed (Participants) | 77
  Day 15 | 23.8 (28.4)
  Day 29: number analyzed (Participants) | 69
  Day 29 | 26.4 (13.7)
  Day 43: number analyzed (Participants) | 69
  Day 43 | 32.3 (35.8)
  Day 57: number analyzed (Participants) | 56
  Day 57 | 32.7 (18.8)
  Day 71: number analyzed (Participants) | 52
  Day 71 | 33.5 (21.1)
  Day 85: number analyzed (Participants) | 42
  Day 85 | 45.5 (53.6)
  Day 99: number analyzed (Participants) | 37
  Day 99 | 40.3 (24.0)
  Day 169: number analyzed (Participants) | 24
  Day 169 | 43.6 (19.6)
  Day 211: number analyzed (Participants) | 1
  Day 211 | 57.2
  Day 253: number analyzed (Participants) | 11
  Day 253 | 38.4 (15.7)
  Day 337: number analyzed (Participants) | 4
  Day 337 | 43.9 (23.7)
  Day 421: number analyzed (Participants) | 2
  Day 421 | 61.4 (7.79)

15. Secondary Outcome: Part B: Interim Analysis: Overall Survival (OS) Time
Description: The OS time was defined as the time from first administration of study treatment until the date of death. OS was calculated using following formula = (date of death - date of the first dose of study treatment + 1)/30.4375 (months).
Time Frame: Up to 161 weeks (Data reported are per pre-specified interim analysis with a data cut-off date of 2 May 2019)
Population: Full Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
Months | 20.3 [0.5 to 34.9]

16. Secondary Outcome: Part B: Final Analysis: Overall Survival (OS) Time
Description: as for outcome 15
Time Frame: Time from first administration of trial treatment until death (Up to 396 weeks)
Population: Full Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
months | 20.3 [0.5 to 65.8]

17. Secondary Outcome: Part B: Number of Participants With Confirmed Best Overall Response (BOR) as Per Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
Description: as for outcome 1
Time Frame: Up to 396 weeks
Population: Full Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
Participants
  Complete Response | 19
  Partial Response | 27
  Stable Disease | 12
  Non-complete Response/ Non-progressive Disease | 1
  Progressive Disease | 48
  Not evaluable | 9

18. Secondary Outcome: Part B: Duration of Response According to Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
Description: The duration of response as determined from IERC tumor assessment was calculated for each participant with a confirmed response (CR or PR) as the time from first observation of response until first observation of documented disease progression or death when death occurs within 12 weeks of the last tumor assessment, whichever occurs first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions.
Time Frame: Up to 396 weeks
Population: Full Analysis Set included all participants who received at least 1 dose of study treatment. Here "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 46
Months | 18.2 [1.2 to 28.3]

19. Secondary Outcome: Part B: Progression-Free Survival (PFS) Time According to Response Evaluation Criteria in Solid Tumors Version (RECIST) 1.1
Description: as for outcome 4
Time Frame: Up to 396 weeks
Population: Full Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Median (Full Range); unit: Months
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
Months | 4.1 [0.03 to 29.6]

20. Secondary Outcome: Part B: Number of Participants With Treatment-Related (TR) Treatment-Emergent Adverse Events (TEAEs), Treatment-Related Serious TEAEs and Treatment-Related TEAEs Leading to Death
Description: as for outcome 5
Time Frame: Up to 396 weeks
Population: Full Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
Participants
  Participants with TR-TEAEs | 94
  Participants with TR-Serious-TEAEs | 17
  Participants with TR-TEAEs leading to Death | 0

21. Secondary Outcome: Part B: Participant's Response Status According to RECIST 1.1 at 6 and 12 Months
Description: as for outcome 11
Time Frame: At Month 6 and 12
Population: Full Analysis Set included all participants who received at least 1 dose of study treatment.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
Percentage of Participants
  In-response at Month 6 | 33.6 [25.1 to 43.0]
  In-response at Month 12 | 26.7 [18.9 to 35.7]
  Not in-response at Month 6 | 66.4
  Not in-response at Month 12 | 73.3

22. Secondary Outcome: Part B: Number of Participants With Positive Treatment Emergent Anti-Avelumab Antibodies
Description: Serum samples were analyzed by a validated electrochemiluminescence immunoassay to detect the presence of antidrug antibodies (ADA). Samples that screened positive were subsequently tested in a confirmatory assay. Those that confirmed positive were titered for a quasi-quantitative result. Number of participants with positive treatment emergent anti-Avelumab antibodies were reported. Participants not positive prior to treatment with avelumab and with at least one positive result in the human-Antihuman Antibodies assay were characterized as treatment-emergent.
Time Frame: Up to 161 weeks
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 110
Participants | 8

23. Secondary Outcome: Part B: Serum Concentration at End of Infusion (CEOI) of Avelumab
Description: Serum concentration at end of infusion (CEOI) of Avelumab is reported.
Time Frame: At Day 1, 43 and 169
Population: PK Analysis Set included all participants who received at least 1 dose of avelumab, and provided at least 1 measurable post-dose concentration. Here "Number analyzed" signifies those participants who were evaluable at specified time-point for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
Microgram per milliliter
  Day 1: number analyzed (Participants) | 104
  Day 1 | 237 (31.1)
  Day 43: number analyzed (Participants) | 78
  Day 43 | 244 (32.1)
  Day 169: number analyzed (Participants) | 41
  Day 169 | 255 (27.7)

24. Secondary Outcome: Part B: Minimum Serum Post-dose (Ctrough) Concentration of Aveluamb
Description: Minimum serum post-dose (Ctrough) concentration of avelumab was reported.
Time Frame: Day 15, Day 29, Day 43, Day 85, Day 127, Day 169, Day 253, Day 337, Day 421, Day 505, Day 589, Day 673
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Microgram per milliliter
Arm/Group | Part B: Avelumab
Number analyzed (Participants) | 116
Microgram per milliliter
  Day 15: number analyzed (Participants) | 100
  Day 15 | 22.2 (57.5)
  Day 29: number analyzed (Participants) | 86
  Day 29 | 27.8 (80.2)
  Day 43: number analyzed (Participants) | 76
  Day 43 | 27.5 (89.4)
  Day 85: number analyzed (Participants) | 61
  Day 85 | 29.4 (130.4)
  Day 127: number analyzed (Participants) | 54
  Day 127 | 37.0 (65.6)
  Day 169: number analyzed (Participants) | 45
  Day 169 | 45.6 (60.3)
  Day 253: number analyzed (Participants) | 47
  Day 253 | 39.9 (53.0)
  Day 337: number analyzed (Participants) | 36
  Day 337 | 39.5 (37.3)
  Day 421: number analyzed (Participants) | 24
  Day 421 | 43.6 (30.3)
  Day 505: number analyzed (Participants) | 14
  Day 505 | 41.8 (30.4)
  Day 589: number analyzed (Participants) | 4
  Day 589 | 57.5 (24.1)
  Day 673: number analyzed (Participants) | 5
  Day 673 | 44.9 (21.4)

ADVERSE EVENTS:
Time Frame: Part A: Up to 325 weeks; Part B: Up to 396 weeks
Description: Adverse events were reported as per MedDRA v21.1 for Part A arm and MedDRA v22.0 for Part B.
Arm/Group | Part A: Avelumab | Part B: Avelumab
All-Cause Mortality (participants affected / at risk) | 63/88 | 72/116
Serious Adverse Events (participants affected / at risk) | 48/88 | 58/116
Other Adverse Events (participants affected / at risk) | 86/88 | 114/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Avelumab (N=88) | Part B: Avelumab (N=116)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Microcytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Eyelid function disorder (Eye disorders) | 1 | 0
Glaucoma (Eye disorders) | 1 | 0
Retinal artery occlusion (Eye disorders) | 1 | 0
Ulcerative keratitis (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 2
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 2 | 1
Oesophageal spasm (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 1 | 2
Chest pain (General disorders) | 1 | 1
Disease progression (General disorders) | 9 | 10
Fatigue (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 2 | 6
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Liver injury (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0
Diabetic foot infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 1
Pneumonia (Infections and infestations) | 1 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 3
Transaminases increased (Investigations) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Bundle branch block right (Cardiac disorders) | 0 | 1
Myocarditis (Cardiac disorders) | 0 | 1
Diplopia (Eye disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Diverticulum (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 2
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Gait disturbance (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Endocarditis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
Infective exacerbation of bronchiectasis (Infections and infestations) | 0 | 1
Peritonitis (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 4
Streptococcal infection (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 1
Radiation skin injury (Injury, poisoning and procedural complications) | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1
Liver function test increased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 1
Post herpetic neuralgia (Nervous system disorders) | 1 | 0
Autoimmune neuropathy (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Paraneoplastic encephalomyelitis (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy in malignant disease (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 4 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 3
Renal impairment (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epiglottic cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 2
Shock haemorrhagic (Vascular disorders) | 0 | 1
Vascular purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Knee arthroplasty (Surgical and medical procedures) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Diabetes insipidus (Endocrine disorders) | 1 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0
Autoimmune colitis (Gastrointestinal disorders) | 1 | 0
Autoimmune disorder (Immune system disorders) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Haematoma infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0
Spinal cord infection (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Intraocular pressure increased (Investigations) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: Avelumab (N=88) | Part B: Avelumab (N=116)
Anaemia (Blood and lymphatic system disorders) | 14 | 19
Lymphopenia (Blood and lymphatic system disorders) | 7 | 9
Eosinophilia (Blood and lymphatic system disorders) | 0 | 6
Abdominal pain (Gastrointestinal disorders) | 11 | 11
Constipation (Gastrointestinal disorders) | 16 | 29
Diarrhoea (Gastrointestinal disorders) | 23 | 18
Nausea (Gastrointestinal disorders) | 24 | 22
Vomiting (Gastrointestinal disorders) | 13 | 10
Asthenia (General disorders) | 10 | 24
Chills (General disorders) | 10 | 14
Fatigue (General disorders) | 34 | 27
Oedema peripheral (General disorders) | 19 | 15
Pyrexia (General disorders) | 9 | 13
Nasopharyngitis (Infections and infestations) | 8 | 8
Upper respiratory tract infection (Infections and infestations) | 6 | 8
Bronchitis (Infections and infestations) | 5 | 7
Infusion related reaction (Injury, poisoning and procedural complications) | 12 | 10
Fall (Injury, poisoning and procedural complications) | 0 | 9
Alanine aminotransferase increased (Investigations) | 7 | 9
Aspartate aminotransferase increased (Investigations) | 7 | 6
Blood bilirubin increased (Investigations) | 0 | 6
Blood creatinine increased (Investigations) | 6 | 10
Blood creatine phosphokinase increased (Investigations) | 7 | 7
Lipase increased (Investigations) | 5 | 10
Weight decreased (Investigations) | 14 | 18
Decreased appetite (Metabolism and nutrition disorders) | 21 | 16
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 7
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 13 | 13
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 0
Dizziness (Nervous system disorders) | 12 | 0
Headache (Nervous system disorders) | 10 | 0
Insomnia (Psychiatric disorders) | 6 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 28
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 16
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 5 | 9
Erythema (Skin and subcutaneous tissue disorders) | 5 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 18
Rash (Skin and subcutaneous tissue disorders) | 13 | 11
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 7
Hypertension (Vascular disorders) | 11 | 11
Hypothyroidism (Endocrine disorders) | 6 | 0
Vision blurred (Eye disorders) | 5 | 0
Cellulitis (Infections and infestations) | 5 | 0
Sinusitis (Infections and infestations) | 5 | 0
Weight increased (Investigations) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 6 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Anxiety (Psychiatric disorders) | 7 | 0
Lymphoedema (Vascular disorders) | 6 | 0
Hypotension (Vascular disorders) | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-25): https://cdn.clinicaltrials.gov/large-docs/47/NCT02155647/Prot_001.pdf
  • Statistical Analysis Plan (2016-03-31): https://cdn.clinicaltrials.gov/large-docs/47/NCT02155647/SAP_000.pdf